CLINICAL TRIAL: NCT06565611
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Clinical Study Investigating the Safety, Tolerability, and Effectiveness of the Co-Administration of Bremelanotide With Tirzepatide (GLP-1/GIP) for the Treatment of Obesity
Brief Title: A Phase 2 Study Evaluating the Co-Administration of Bremelanotide With Tirzepatide for the Treatment of Obesity
Acronym: BMT-801
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMT-801
Record Dates: First submitted 2024-06-05; First posted 2024-08-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Obesity; Tirzepatide; Bremelanotide; BMI
MeSH Terms: conditions — Obesity | interventions — bremelanotide; Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- tirzepatide and bremelanotide Combination Therapy (Active Comparator)
  Interventions: Drug: bremelanotide; Drug: tirzepatide
- tirzepatide Monotherapy (Placebo Comparator): N=1
  Interventions: Drug: tirzepatide
- bremelanotide Monotherapy (Placebo Comparator)
  Interventions: Drug: bremelanotide
- Placebo (No Intervention)

INTERVENTIONS:
Drug: bremelanotide — bremelanotide (BMT) sterile aqueous solution for subcutaneous injection, provided as autoinjectors containing 0.3 mL volume
  Arms: bremelanotide Monotherapy; tirzepatide and bremelanotide Combination Therapy
Drug: tirzepatide — tirzepatide (GLP-1/GIP) will be provided in its commercial form for SC injection.
  Arms: tirzepatide Monotherapy; tirzepatide and bremelanotide Combination Therapy

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled study designed to assess the safety and efficacy of bremelanotide (BMT) used in combination with tirzepatide therapy in the treatment of obesity in subjects with a BMI ranging from 30.0 to 45.0 kg/m2 (inclusive).

DETAILED DESCRIPTION:
A total of approximately 108 subjects at approximately five (5) centers within the United States (US), will be enrolled into the study for 8 weeks of treatment. Subjects who provide written informed consent and meet all initial eligibility criteria will enter into Screening. The subjects' historical and current medical data will be collected, reviewed, and recorded to be used as baseline values.

Enrolled subjects will begin the study and go through 2 treatment periods:

* "Treatment Period 1" - 4 weeks of tirzepatide therapy only
* "Treatment Period 2" - 4 weeks of combination therapy of bremelanotide, Placebo, or tirzepatide therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged between 18-65 years of age, inclusive at the time of consent.
2. Have a body mass index (BMI) of 30.0 to 45.0 kg/m^2 (inclusive) at screening.
3. Female subjects must have a negative urine pregnancy test at screening, if of childbearing potential or be of non-childbearing potential. If the urine test is positive or cannot be confirmed as negative, then the subject must have a negative serum pregnancy test (hCG). Non-childbearing potential is defined as (by other than medical reasons):

   1. Age ≥ 50 years, no menses for at least one year, per subject self-report.
   2. Documented hysterectomy, bilateral tubal ligation, or bilateral oophorectomy.
4. For female subjects who are Women of childbearing potential (WOCBP), subject must agree to abstain from heterosexual intercourse or use a highly effective contraceptive(s) (with a failure rate of <1% per year), as described in the protocol, during the treatment and follow-up and for at least 90 days after the last dose of bremelanotide. Hormonal-based contraception is to be employed for a minimum of 28 days prior to Day 0. Oral hormonal contraceptives should be combined estrogen and progesterone. If a progesterone-only oral contraceptive is used, then a second method of birth control should be used as well. Acceptable forms of contraception include:

   * Surgical sterilization of the subject or male partner;
   * FDA- or Health Canada-approved female hormonal contraceptives;
   * An IUD;
   * Essure® (transcervical sterilization);
   * "Double-barrier" contraception defined as:

     * condom + spermicide, or
     * condom + diaphragm (which is used with a spermicide).
5. Female subjects must agree not to donate eggs (ova, oocytes) for any purpose during the treatment and follow-up and for at least 30 days after the last dose of BMT.
6. Male subjects must agree to abstain from heterosexual intercourse or use double barrier protection with condom and spermicide with any WOCBP sexual partner from screening and continuing for at least 30 days after the last dose of BMT:

   a. Alternatively, documented sterilization confirmed by the absence of sperm in the ejaculate or ≥ one-year post-operative from vasectomy.
7. Male subjects must agree not to donate sperm for at least 30 days after the last dose of BMT.
8. Subjects must be willing to self-inject.
9. Subjects must have the ability to complete the study in compliance with the protocol and all instructions.
10. Subjects must have the ability to understand and provide written informed consent.

Exclusion Criteria:

1. Females who are pregnant, breastfeeding or plan to become pregnant.
2. Have a known allergy or intolerance to Melanocortin peptides.
3. Subjects with a positive Serum Antigen/Antibody Hepatitis Panel (Hep B and C) and HIV antibody test Human Immunodeficiency Virus (HIV) antibody.

   Note: subject with positive hepatitis C antibody but negative PCR test for active Hepatitis C viral shedding will be allowed to participate in the study. Subjects with a positive Hepatitis B surface antigen antibody or core antigen antibody will be allowed to participate in the study. Subjects with circulating hepatitis B surface antigen or have a positive PCR test for active hepatitis B virus will NOT be allowed to participate in the study.
4. Subjects with active alcohol dependence and/or drug use (with Cannabis exception) as assessed by the Investigator will be excluded from the study.
5. Have significant medical illnesses that cannot be adequately controlled with appropriate therapy and may obscure toxicity, dangerously alter drug metabolism, or compromise the subject's ability to participate in the trial, as determined by the Investigator, such as endocrinologic disorders accounting for obesity such as Cushing Disease, syndrome or monogenic obesity and exclusions of organ transplant recipients, those on wait lists, or those on anti-rejection medication as the potential effect on gastric emptying effecting pharmacokinetics.
6. Has been on bremelanotide therapy (Vyleesi) within the past 6 months prior to screening date.
7. Within the past three month, has used cyclosporine A, adrenocorticotropic hormones, long-term corticosteroids (> 20 mg qd or its equivalent for > 3 months), or cytotoxic agents.
8. Has had clinically significant body weight change (≥5%) or dieting attempts in the prior 90 days (per subject reported information) and Treatment Period 1.
9. Use of Anti-Obesity Medication (AOM) within a 90-day period prior to screening (Note: subjects who have taken or are still taking tirzepatide may participate in study if exclusion criteria #8 has not been met. AOM medications will also include medications that are being used off-label for weight loss).
10. Prior obesity or weight loss surgery or presence of gastrointestinal implant or bariatric surgery or other weight loss procedures within 2 years of screening (i.e. liposuction, abdominoplasty, intragastric balloon, cholecystectomy, etc.)
11. Has HbA1c ≥ 6.5 % or fasting glucose ≥126.0 mg/dL. (either test can be used to establish eligibility).
12. Has type 1 diabetes.
13. Has taken any experimental drug or therapy within 28 days / 5 half-lives of trial treatment or concurrently participating in another clinical trial.
14. Has a history of clinically significant bradycardia and/or a heart rate less than 50 bpm at screening.
15. Has multiple endocrine neoplasia syndrome type 2.
16. Plan for blood donations during the study and within 30 days following completion of or early discontinuation from the trial.
17. Planned bariatric surgery or planned major surgeries during the study time period.
18. Has personal or family history of MEN 2 syndromes or Medullary Thyroid Cancer.
19. Prior hypersensitivity to tirzepatide component.
20. Has hypertension (by medical history or by screening vital signs) and/or known cardiovascular disease.

    Note: If subject presents at screening with elevated blood pressure and no supporting evidence of hypertension; subject may wait approximately 1 hour to have blood pressure rechecked; if readings are still elevated, subject may return to the site approximately 24 hours later to have blood pressure rechecked.
21. Is taking concomitant oral drugs that are dependent on threshold concentrations for efficacy (e.g., antibiotics) since bremelanotide slows gastric emptying and thus has the potential to reduce the rate and extent of absorption of concomitantly administered oral medications
22. Has a diagnosis of type 2 diabetes
23. Has Clinically significant ECG abnormalities on ECG at Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in body weight between treatment arms | Change from the baseline (Visit 2/Day 1) to Visit 10 (Day 57)
  Percent change in patient weight from baseline (Visit 2/Day 1) to Visit 10 (Day 57) for the BMT/tirzepatide combination group compared to placebo

OTHER OUTCOMES:
Change in Body Weight | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) in body weight (lbs.) between treatment arms
Change in Overall Appetite Suppression | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint is the change from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) in overall appetite suppression, as quantified by the Visual Analog Scale (VAS), between treatment arms. The Hunger and Satiety Visual Analogue Scales (VAS) yields a composite score ranging from 0 to 100, where 0 represents extreme hunger and 100 represents complete satiety. A higher VAS composite score indicates greater appetite suppression efficacy of the treatment.
Change in Appetite Suppression Subscales | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint assesses the change from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) in individual appetite suppression subscales (hunger, fullness, satiety, and prospective food consumption) between treatment arms. The Hunger and Satiety Visual Analogue Scales (VAS) comprise four distinct subscales, each quantifying specific aspects of appetite suppression: hunger, fullness, satiety, and prospective food consumption. These subscales permit independent assessment.
  * The hunger subscale, ranging from 0 to 100, quantifies subjective hunger, where 0 indicates minimal hunger and 100 maximal hunger. A score of 0 denotes optimal efficacy.
  * The fullness subscale, ranging from 0 to 100, quantifies subjective fullness, where 0 signifies absence of fullness and 100 complete fullness. A score of 100 denotes optimal efficacy.
  * The satiety subscale, ranging from 0 to 100, quantifies subjective satiety, where 0 signifies complete emptiness and 100 comp
Change in Percent Body Fat | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) in percent body fat between treatment arms
Change in BMI | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) in BMI between treatment arms
Change in Skeletal Muscle Mass | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the change in skeletal muscle mass from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) between treatment arms. Skeletal muscle mass is quantified utilizing Bioelectrical Impedance Analysis (BIA) as the measurement modality. It is acknowledged that the observed range of skeletal muscle mass values is subject to inter-individual variability, influenced by factors including, but not limited to, age, gender, hydration status, recent dietary intake, and body temperature. Skeletal muscle mass assessment will be conducted in conjunction with the analysis of percent body fat and visceral fat level to provide a comprehensive evaluation of lean tissue composition.
Change in Visceral Fat Level | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the change in visceral fat level from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) between treatment arms. Visceral fat is quantified utilizing Bioelectrical Impedance Analysis (BIA) as the measurement modality. It is acknowledged that the observed range of visceral fat values is subject to inter-individual variability, influenced by factors including, but not limited to, age, gender, hydration status, recent dietary intake, and body temperature. A visceral fat assessment will be conducted in conjunction with the analysis of percent body fat and skeletal muscle mass to provide a comprehensive evaluation of lean tissue composition.
Number of participants with abnormal laboratory tests results | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the incidence of participants exhibiting clinically significant changes in laboratory test results from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57), specifically focusing on deviations from reference ranges within the comprehensive metabolic panel (CMP) and lipid panel, between treatment arms.
Change in Neck and Waist Measurements | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the change in neck and waist circumferences from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) between treatment arms. Circumferential measurements are obtained utilizing a calibrated tape measure with an imperial scale (inches). Neck circumference is determined by measuring the horizontal circumference at the level of the larynx. Waist circumference is assessed at the umbilicus in male participants, and at the midpoint between the inferior border of the sternum and the umbilicus in female participants. In female participants, hip circumference is additionally measured at the level of maximum gluteal protrusion.
Change in IIEF Domain Score | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the change in the International Index of Erectile Function (IIEF) Erectile Function (EF) domain score from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) between treatment arms. The IIEF questionnaire, utilized for this assessment, yields an EF domain score ranging from 6 to 30, with higher scores indicative of improved erectile function.
Change in EDQ Score | Change from the Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57)
  This exploratory endpoint evaluates the change in the Elements of Desire Questionnaire (EDQ) total score from Visit 2 baseline and Treatment Period 2 baseline (Day 29) to Visit 10 (Day 57) between treatment arms. The Elements of Desire Questionnaire (EDQ) is the instrument employed for this assessment. The total score is derived from the mean of the nine EDQ items, each rated on a scale of 1 to 5, where 5 represents the maximum level of desire and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jordan, Study Director — Palatin
Locations (4):
- United States (4):
  - University Clinical Research-DeLand LLC, d/b/a Accel Research, DeLand, Florida
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Lynn Institute of Chattanooga, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No